CLINICAL TRIAL: NCT01634295
Title: A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of a Fixed Dose Combination of S-Amlodipine and Telmisartan(CKD-828) Versus S-Amlodipine Monotherapy in Patients With Stage 2 Hypertension
Brief Title: Efficacy and Safety of CKD-828 to Stage 2 Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 130HT11P
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Hypertension
Keywords: CKD-828; Hypertension; Stage 2 Hypertension; S-Amlodipine; Telmisartan
MeSH Terms: conditions — Hypertension | interventions — levamlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-828 2.5/40, 2.5/80, 5/80mg (Experimental)
  Interventions: Drug: CKD-828 2.5/40mg; Drug: CKD-828 5/40mg; Drug: CKD-828 5/80mg
- S-Amlodipine 2.5, 5mg (Active Comparator)
  Interventions: Drug: S-amlodipine 2.5mg; Drug: S-amlodipine 5mg

INTERVENTIONS:
Drug: CKD-828 2.5/40mg — * Fixed dose combination of S-amlodipine 2.5mg and Telmisartan 40mg QD 2 weeks.
  * With the others investigation product placebo 4 tabs QD 2 weeks.
  Other Names: CKD-828
  Arms: CKD-828 2.5/40, 2.5/80, 5/80mg
Drug: CKD-828 5/40mg — * Fixed dose combination of S-amlodipine 5mg and Telmisartan 40mg QD 2 weeks.
  * With the others investigation product placebo 4 tabs QD 2 weeks.
  Other Names: CKD-828
  Arms: CKD-828 2.5/40, 2.5/80, 5/80mg
Drug: CKD-828 5/80mg — * Fixed dose combination of S-amlodipine 5mg and Telmisartan 80mg QD 6 weeks.
  * With the others investigation product placebo 4 tabs QD 6 weeks.
  Other Names: CKD-828
  Arms: CKD-828 2.5/40, 2.5/80, 5/80mg
Drug: S-amlodipine 2.5mg — * S-amlodipine 2.5mg QD 4 weeks
  * With the others investigation product placebo 4 tabs QD 4 weeks.
  Other Names: Anydipine S
  Arms: S-Amlodipine 2.5, 5mg
Drug: S-amlodipine 5mg — * S-amlodipine 2.5mg QD 6weeks
  * With the others investigation product placebo 4 tabs QD 6 weeks.
  Other Names: Anydipine S
  Arms: S-Amlodipine 2.5, 5mg

SUMMARY:
The aim of present study is to evaluate the efficacy and safety of two dose combination of S-Amlodipine/Telmisartan (2.5/40mg, 2.5/80mg and 5/80mg) compared with S-Amlodipine monotherapy (2.5mg and 5mg) in patients with Stage 2 hypertension.

DETAILED DESCRIPTION:
* In patients with Stage 2 hypertension to determine the efficacy and safety of S-Amlodipine/Telmisartan (2.5/40mg, 2.5/80mg and 5/80mg) or S-Amlodipine monotherapy (2.5mg and 5mg) during 10 weeks.
* This study is consist of placebo run-in period(2 weeks_single blind) and treatment period(10 weeks_double blind.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* at the screening visit

  * antihypertensive drugs not taking: 160mmHg ≤ sitSBP < 200mmHg
  * antihypertensive drugs taking: 140mmHg ≤ sitSBP < 180mmHg
* at the randomization visit(160mmHg ≤ sitSBP < 200mmHg)
* willing and able to provide written informed consent

Exclusion Criteria:

* mean sitting DBP ≥ 120mmHg or mean sitting SBP ≥ 200mmHg at the screening visit and randomization visit
* for the past four weeks based on beginning of administration, patients took over four antihypertensive drugs
* known or suspected secondary hypertension(ex. aortic coarctation, Primary hyperaldosteronism, renal artery stenosis, pheochromocytoma)
* has severe heart disease(Heart failure NYHA functional class 3, 4), ischaemic heart diseasesstatus need to treatment, myocardiopathy, Valve disease, arrhythmia and so on and operated Coronary angioplasty
* has cerebrovascular disease as cerebral infarction, cerebral hemorrhage within 6 months
* Type I Diabetes Mellitus, Type II Diabetes Mellitus with poor glucose control as defined by fasting glucosylated hemoglobin(HbA1c) > 8%)
* known severe or malignant retinopathy
* defined by the following laboratory parameters:

  * hepatic dysfunction(AST/ALT > UNL X 3)
  * renal dysfunction(serum creatinine > UNL X 1.5)
  * hypopotassemia(K < 3.0mmol/L) or hyperpotassemia (K>5.5 mmol/L)
* acute or chronic inflammatory status need to treatment
* need to additional antihypertensive drugs during the study
* need to concomitant medications known to affect blood pressure during the study
* history of angioedema related to ACE inhibitors or Angiotensin II Receptor Blockers
* known hypersensitivity related to either study drug
* history of drug or alcohol dependency within 6 months
* any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of investigational products(ex. gastrointestinal tract surgery such as gastrectomy, gastroenterostomy or bypass, active inflammatory bowel syndrome within 12 months prior to screening, gastric ulcers need to treatment, gastrointestinal/rectal bleeding, impaired pancreatic function such as pancreatitis, obstructions of the urinary tract or difficulty in voiding)
* administration of other study drugs within 4weeks prior to randomization
* premenopausal women(last menstruation < 1year) not using adequate contraception, pregnant or breast-feeding
* history of malignancy including leukemia and lymphoma within the past 5 years
* in investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mean Sitting systolic Blood Pressure (MSSBP) | After 10 weeks of treatment

SECONDARY OUTCOMES:
Mean Sitting systolic Blood Pressure (MSSBP) | After 2 weeks, 4 weeks and 6 weeks of treatment
Mean Sitting diastolic Blood Pressure (MSDBP) | After 2weeks, 4weeks, 6weeks and 10 weeks of treatment
Control Rate | After 10 weeks of treatment
  Sitting SBP<140mmHg, Sitting DBP<90mmHg
Response Rate | After 10 weeks of treatment
  Reduction of Sitting SBP≥20mmHg, Sitting DBP ≥10mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Tae-hoon An, Ph.D, Principal Investigator — Gachon University Gil Medical Center; Eun-joo Jo, Ph.D, Principal Investigator — The Catholic university of Korea St. Paul's Hospitial; Jong-jin Kim, Ph.D, Principal Investigator — Kyung Hee university Hosipital at Gangdong; Jang-ho Bae, Ph.D, Principal Investigator — Konyang University Hosipital; Chang-kyu Park, Ph.D, Principal Investigator — Korea University Guro Hospital; Young-dae Kim, Ph.D, Principal Investigator — Dong-A University; Chul-ho Kim, Ph.D, Study Chair — Seoul National University Bundang Hospital; Sae-Joong Lim, Ph.D, Principal Investigator — Gangnam Severance Hospital; Uk-Bum Phyun, Ph.D, Principal Investigator — Ewha Women University Mokdong Hospital; Gyu-Rok Han, Ph.D, Principal Investigator — Kangdong Sacred Heart Hospital; Sang Hyun Kim, Ph.D, Principal Investigator — Seoul National University Boramae Hospital
Locations (1):
- Seoul national university Bundang Hospital, Bundang-gu, Gyeonggi-do, South Korea